CLINICAL TRIAL: NCT00431171
Title: A Three Month, Open-label, Single-arm Trial Evaluating the Safety and Pharmacokinetics of Oral Lithium in Patients Diagnosed With Chronic Spinal Cord Injury
Brief Title: Safety and Pharmacokinetics Study of Oral Lithium in Patients With Chronic Spinal Cord Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: China Spinal Cord Injury Network (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN101
Record Dates: First submitted 2007-02-01; First posted 2007-02-05 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injuries; lithium
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Lithium Carbonate

INTERVENTIONS:
Drug: Lithium carbonate

SUMMARY:
The current study is a phase I open-label clinical trial to examine plasma levels after oral lithium treatments in 20 subjects with chronic spinal cord injury. The subjects will receive standard doses of oral lithium used in treatment of manic depression. The goal of the trial is to show feasibility and safety of maintaining plasma levels of 0.6 mmol/L to 1.2 mmol/L for six weeks in subjects with chronic spinal cord injury.

DETAILED DESCRIPTION:
Patients with spinal cord injury (SCI) usually have permanent and often devastating neurological deficits and disability. There has been successful research in a number of fields that may someday help people with spinal cord injuries.

The planned treatment trials will focus on the effects of oral lithium on neurological function in people with chronic spinal cord injury and those that have received umbilical cord blood mononuclear cell transplants to the spinal cord. The interest in these two treatments derives from recent reports indicating that umbilical cord blood stem cells may be beneficial for spinal cord injury and that lithium may promote regeneration and recovery of function after spinal cord injury. Both lithium and umbilical cord blood are widely available therapies that have long been used to treat diseases in humans.

The current study is a phase I open-label clinical trial to examine plasma levels after oral lithium treatments in 20 subjects with chronic spinal cord injury. The subjects will receive standard doses of oral lithium used in treatment of manic depression. The goal of the trial is to show feasibility and safety of maintaining plasma levels of 0.6 mmol/L to 1.2 mmol/L for six weeks in subjects with chronic spinal cord injury.

Lithium attracted much attention as a potential neuroregenerative therapy based on experiments in animal models of SCI in 2004. However, toxic levels of lithium (>1.5 mmol/L) are close to the effective levels (0.6 - 1.2 mmol/L). At toxic levels, patients may become confused and lethargic, have diarrhea, upset stomach, and develop tremors, ataxia, dysarthria, and nystagmus. Lithium toxicity may be compounded by sodium depletion or diuretics (thiazides) that inhibit kidney sodium upgrade and ACE inhibitors. Plasma levels also depend on fluid input/output. Therefore, care will be taken to titrate the dose and to test plasma levels of the drug at the beginning, at day 2, 7, and week 6 during the treatment period.

Acute toxicity usually produces relatively mild symptoms. Chronic lithium toxicity may lead to more severe neurotoxic symptoms. However, these symptoms usually develop after 3-5 years of treatment.

Data obtained from this study will be used to develop future chronic spinal cord injury clinical studies: (1) randomized controlled trials with lithium versus placebo; and (2) randomized controlled trials comparing effects of lithium and placebo on subjects who have received umbilical cord blood mononuclear cell transplants to the spinal cord.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender and 18 - 60 years of age (preferably 10 males and females each)
* Subjects with chronic spinal cord injury (defined as 12 months or more post spinal cord injury), as confirmed by a MRI
* Subjects with neurological status: ASIA A, B or C
* Subjects must be able to read, understand, and complete the VAS
* Subjects who have voluntarily signed* and dated* an informed consent form, approved by an IEC/IRB, prior to any study-specific procedures *If a subject consents to participation but is not in a position to personally sign and date the informed consent form because of his or her physical condition, the consent must be confirmed at the time of consent orally, signed on behalf by the subject's relative, and by an impartial witness who is present throughout the whole informed consent process.

Exclusion Criteria: Subjects are excluded if they have

* a history of hypersensitivity to lithium
* significant renal, cardiovascular, hepatic and psychiatric diseases
* significant medical diseases or infection
* brain injury
* Addison's disease
* debilitation or dehydration
* recently taken or are taking diuretics or other drugs with known interaction with lithium, such as tricyclic antidepressants, NSAIDs and tetracycline
* a history of alcohol abuse or drug abuse, or if they are
* pregnant or lactating women;
* female of childbearing potential and are unwilling to use an effective contraceptive method while enrolled in the study;
* subjects who are currently participating in another investigational study or have been taking any investigational drug within the last 4 weeks prior to screening of this study (Visit 1); and finally,
* any criteria, which, in the opinion of the investigator, suggest that the subject would not be compliant with the study protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Incidence of clinical adverse events including known and unknown adverse events, and changes from baseline in vital signs, ECGs and laboratory parameters

SECONDARY OUTCOMES:
Plasma lithium level

CONTACTS AND LOCATIONS:
Overall Officials: Yat-wa Wong, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- MacLehose Medical Rehabilitation Centre, Pokfulam, Hong Kong SAR, China

REFERENCES:
- [Background] Yick LW, So KF, Cheung PT, Wu WT. Lithium chloride reinforces the regeneration-promoting effect of chondroitinase ABC on rubrospinal neurons after spinal cord injury. J Neurotrauma. 2004 Jul;21(7):932-43. doi: 10.1089/neu.2004.21.932. PMID 15307905
- [Background] Phiel CJ, Klein PS. Molecular targets of lithium action. Annu Rev Pharmacol Toxicol. 2001;41:789-813. doi: 10.1146/annurev.pharmtox.41.1.789. PMID 11264477
- [Background] Etheridge SL, Spencer GJ, Heath DJ, Genever PG. Expression profiling and functional analysis of wnt signaling mechanisms in mesenchymal stem cells. Stem Cells. 2004;22(5):849-60. doi: 10.1634/stemcells.22-5-849. PMID 15342948
- [Background] Merendino RA, Arena A, Gangemi S, Ruello A, Losi E, Bene A, D'Ambrosio FP. In vitro interleukin-8 production by monocytes treated with lithium chloride from breast cancer patients. Tumori. 2000 Mar-Apr;86(2):149-52. doi: 10.1177/030089160008600208. PMID 10855853
- [Background] Merendino RA, Arena A, Gangemi S, Ruello A, Losi E, Bene A, Valenti A, D'Ambrosio FP. In vitro effect of lithium chloride on interleukin-15 production by monocytes from IL-breast cancer patients. J Chemother. 2000 Jun;12(3):252-7. doi: 10.1179/joc.2000.12.3.252. PMID 10877522
- [Background] Merendino RA, Mancuso G, Tomasello F, Gazzara D, Cusumano V, Chillemi S, Spadaro P, Mesiti M. Effects of lithium carbonate on cytokine production in patients affected by breast cancer. J Biol Regul Homeost Agents. 1994 Jul-Sep;8(3):88-91. PMID 7754794
- [Background] De Boer J, Wang HJ, Van Blitterswijk C. Effects of Wnt signaling on proliferation and differentiation of human mesenchymal stem cells. Tissue Eng. 2004 Mar-Apr;10(3-4):393-401. doi: 10.1089/107632704323061753. PMID 15165456
- [Background] de Boer J, Siddappa R, Gaspar C, van Apeldoorn A, Fodde R, van Blitterswijk C. Wnt signaling inhibits osteogenic differentiation of human mesenchymal stem cells. Bone. 2004 May;34(5):818-26. doi: 10.1016/j.bone.2004.01.016. PMID 15121013
- [Background] Ohteki T, Parsons M, Zakarian A, Jones RG, Nguyen LT, Woodgett JR, Ohashi PS. Negative regulation of T cell proliferation and interleukin 2 production by the serine threonine kinase GSK-3. J Exp Med. 2000 Jul 3;192(1):99-104. doi: 10.1084/jem.192.1.99. PMID 10880530
- [Background] Kim JS, Chang MY, Yu IT, Kim JH, Lee SH, Lee YS, Son H. Lithium selectively increases neuronal differentiation of hippocampal neural progenitor cells both in vitro and in vivo. J Neurochem. 2004 Apr;89(2):324-36. doi: 10.1046/j.1471-4159.2004.02329.x. PMID 15056276
- [Background] Aubert J, Dunstan H, Chambers I, Smith A. Functional gene screening in embryonic stem cells implicates Wnt antagonism in neural differentiation. Nat Biotechnol. 2002 Dec;20(12):1240-5. doi: 10.1038/nbt763. Epub 2002 Nov 25. PMID 12447396
- [Background] Hellweg R, Lang UE, Nagel M, Baumgartner A. Subchronic treatment with lithium increases nerve growth factor content in distinct brain regions of adult rats. Mol Psychiatry. 2002;7(6):604-8. doi: 10.1038/sj.mp.4001042. PMID 12140783
- [Background] Angelucci F, Mathe AA, Aloe L. Neurotrophic factors and CNS disorders: findings in rodent models of depression and schizophrenia. Prog Brain Res. 2004;146:151-65. doi: 10.1016/s0079-6123(03)46011-1. PMID 14699963
- [Background] Shimomura A, Nomura R, Senda T. Lithium inhibits apoptosis of mouse neural progenitor cells. Neuroreport. 2003 Oct 6;14(14):1779-82. doi: 10.1097/00001756-200310060-00004. PMID 14534419
- [Background] Hashimoto R, Senatorov V, Kanai H, Leeds P, Chuang DM. Lithium stimulates progenitor proliferation in cultured brain neurons. Neuroscience. 2003;117(1):55-61. doi: 10.1016/s0306-4522(02)00577-8. PMID 12605892
- [Background] Willing AE, Zigova T, Milliken M, Poulos S, Saporta S, McGrogan M, Snable G, Sanberg PR. Lithium exposure enhances survival of NT2N cells (hNT neurons) in the hemiparkinsonian rat. Eur J Neurosci. 2002 Dec;16(12):2271-8. doi: 10.1046/j.1460-9568.2002.02300.x. PMID 12492421
- [Background] Mignat C, Unger T. ACE inhibitors. Drug interactions of clinical significance. Drug Saf. 1995 May;12(5):334-47. doi: 10.2165/00002018-199512050-00005. PMID 7669262
- [Background] Chen KP, Shen WW, Lu ML. Implication of serum concentration monitoring in patients with lithium intoxication. Psychiatry Clin Neurosci. 2004 Feb;58(1):25-9. doi: 10.1111/j.1440-1819.2004.01188.x. PMID 14678453
- [Background] Oakley PW, Whyte IM, Carter GL. Lithium toxicity: an iatrogenic problem in susceptible individuals. Aust N Z J Psychiatry. 2001 Dec;35(6):833-40. doi: 10.1046/j.1440-1614.2001.00963.x. PMID 11990895
- [Background] Gitlin M. Lithium and the kidney: an updated review. Drug Saf. 1999 Mar;20(3):231-43. doi: 10.2165/00002018-199920030-00004. PMID 10221853
- [Background] Grignon S, Bruguerolle B. Cerebellar lithium toxicity: a review of recent literature and tentative pathophysiology. Therapie. 1996 Mar-Apr;51(2):101-6. PMID 8763043
- [Background] Kilts CD. The ups and downs of oral lithium dosing. J Clin Psychiatry. 1998;59 Suppl 6:21-6; discussion 27. PMID 9674933
- [Background] Karch FE, Lasagna L. Adverse drug reactions. A critical review. JAMA. 1975 Dec 22;234(12):1236-41. PMID 1242749
- See also: The results of the the captioned study was published in Spinal Cord (2011) ,49 issue — http://www.nature.com/sc/journal/v49/n1/full/sc201069a.html